CLINICAL TRIAL: NCT01222949
Title: A Phase I, Pharmacokinetic Trial, in Healthy Asian and Caucasian Volunteers for Investigating the Pharmacokinetic Profiles of Eurartesim™ (40 mg Dihydroartemisinin (DHA)/320 mg Piperaquine (PQ) Phosphate.
Brief Title: A Pharmacokinetic (PK) Trial in Healthy Asian and Caucasian Volunteers Investigating the PK Profile of Eurartesim™
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Giovanni Valentini, MD, Medical Department, R&D Division, Sigma-Tau ifr SpA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST3073/ST3074-DM09-007
Record Dates: First submitted 2010-10-11; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asian Healthy Volunteers (Experimental): Asian males with a body weight ≤ 65 kg (12 subjects) Asian females with a body weight ≤ 65 kg (12 subjects)
  Interventions: Drug: Eurartesim
- Caucasian Healthy Volunteers (Experimental): Caucasian males with a body weight ≤ 65 kg (12 subjects) Caucasian females with a body weight ≤ 65 kg (12 subjects) Caucasian males with a body weight > 65 kg (24 subjects)
  Interventions: Drug: Eurartesim

INTERVENTIONS:
Drug: Eurartesim — Tablet containing 40 mg of Dihydroartemisinin (DHA) and 320 mg of Piperaquine phosphate (PQP). 3 Tablets a Day for body weight comprised between 36 and 75 kg, 4 tablets for body weight above 75 kg.

SUMMARY:
The Study was designed to evaluate the pharmacokinetics of DHA and PQ in healthy volunteers and to assess the effect of ethnicity (Asian vs Caucasian), gender and body weight on the relative bioavailability of DHA and PQ.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or Asian healthy subjects, Male or female, aged between 18 and 50 years (inclusive)
* Body Mass Index (BMI) between 19.0 kg/m2 and 27.0 kg/m2 inclusive, with a minimum body weight of 36 kg.
* Agreed to use two approved methods of contraception
* Had given written informed consent to participate in this study in accordance with local regulations

Exclusion Criteria:

* Had received or was anticipated to receive a prescription medication within 14 days prior to the start of dosing
* Pregnant or lactating (females only)
* Abnormal laboratory test results deemed clinically significant at screening
* Positive urine drug test or alcohol breath test
* Acute therapy for a serious infection within 30 days of study entry
* History of significant drug allergies or significant allergic reactions
* Had participated in a clinical trial or had received an experimental therapy within 30 days or 10 half-lives of the drug
* Receipt of blood or blood products, or loss or donation of 450 mL or more of blood within 90 days before the first dose administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
PK: tmax, Cmax, AUC0-12(DHA), AUC0-24(PQ), AUC0-inf, λz, t1/2 | During the first and last day of drug administration (day 0 and 2) and followed up till Day 90
  DHA evaluation: At pre-dose on day Day 0 and Day 2 and then at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose.
  PQ evaluation: At pre-dose Day 0 and then at 1, 2, 3, 4, 5, 6, 8, 12, and 16 hours post-dose; then at pre-dose Day 1 and Day 2 and finally at 1, 2, 3, 4, 5, 6, 8, 12, and 16 hours post-dose on day 2; on Day 3, 4, 5, 7, 14, 21, 28, 42, 56 and 90.

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | From Day 0 till Day 90
  Number of TEAEs and number of Subjects experiencing Adverse Events during all the study period
Hematology and blood chemistry changes respect to baseline values | Day 0, Day 3, Day 28, Day 90
  Abnormalities in hematology (Haemoglobin, Hematocrit,RBC count, White cell count and differential count, Platelets) and clinical chemistry (Protein, Sodium, Potassium, Chloride ,Total Bilirubin, Conjugated Bilirubin, Alanine Aminotransferase, Aspartate Aminotransferase, Total Cholesterol, Glucose, Bicarbonate, Urea, Urate, Lactate Dehydrogenase, Albumin, Globulins, Triglycerides, Creatinine, Alkaline Phosphatase, Gamma glutamyltransferase, Total Calcium, Phosphate, C-reactive protein) will be recorded the day of the last study drug intake and after 30 days from the start of the drug treatment
QTc interval prolongation | Day 0, day 3, day 28, day 90
  ECG recordings will be obtained at baseline, after the last drug intake and 30 days follow-up to investigate changes in ECG parameters, and specifically QTc interval changes respect to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - CMAX, a division of IDT Australia Limited, Adelaide
  - Nucleus Network Limited, Melbourne